CLINICAL TRIAL: NCT04469140
Title: Non Exudative Age-Related Macular Degeneration Imaged With Swept Source Optical Coherence Tomography: The Extension Study
Brief Title: Non Exudative AMD Imaged With SS-OCT- Extension
Acronym: BIRC-02
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Image Reading Center (Industry)
Responsible Party: Sponsor
Other Study IDs: BIRC-02 IMPACT SWAGGER
Record Dates: First submitted 2020-06-23; First posted 2020-07-13 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Dry Macular Degeneration
Keywords: AMD; Early AMD; Intermediate AMD; Geographic Atrophy; Nascent GA
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At baseline or follow up, an optional blood sample for future exploratory genetics analysis will be collected if not already collected during the BIRC-01 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cohort 1 'IMPACT Cohort': Subjects with intermediate AMD in both eyes, and at least one eye with a drusen volume in the central 3 mm circle centered on the fovea of at least 0.02mm3 in the absence of GA or nGA as diagnosed with OCT en face imaging OR subjects with AMD (early or intermediate) diagnosed in one eye and exudative AMD diagnosed in the fellow eye will undergo SS-OCT imaging every 3 months for 2 years
  Interventions: Device: SS-OCT imaging
- Cohort 2 'SWAGGER Cohort': Subjects with GA or nGA secondary to AMD that is at least the size of a large druse (125 microns in diameter; 0.05 mm2) and no greater than 7 disc areas (17 mm2) in at least one eye will undergo SS-OCT imaging every 3 months for 2 years
  Interventions: Device: SS-OCT imaging
- Cohort 3: Subjects with GA enrolled in another trial
  Interventions: Device: SS-OCT imaging

INTERVENTIONS:
Device: SS-OCT imaging — All subjects will undergo retinal imaging using the Zeiss PlexElite SS-OCT, a non-contact, non-invasive ocular imaging instrument
  Other Names: Zeiss PlexElite; PlexElite 9000; Swept Source OCT; Optical Coherence Tomography Angiography

SUMMARY:
The investigators wish to better understand the role of the choriocapillaris (CC) in the formation and progression of non-exudative in age related macular degeneration (armd) by imaging the retinal pigment epithelium (rpe) and the choroidal microvasculature and by studying their inter-dependence to determine if the loss of the CC could prove useful as an anatomic clinical trial endpoint in future drug trials.

DETAILED DESCRIPTION:
The investigators wish to better understand the role of the choriocapillaris (CC) in the formation and progression of non-exudative in age related macular degeneration (armd) by imaging the retinal pigment epithelium (rpe) and the choroidal microvasculature and by studying their inter-dependence to determine if the loss of the CC could prove useful as an anatomic clinical trial endpoint in future drug trials. This is an extension of a currently ongoing longitudinal observational study (BIRC-01) (NCT03688243).

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in and completion of the BIRC-01 study
* Clinic diagnosis of non-exudative iAMD in at least one eye with a drusen volume in the central 3 mm circle centered on the fovea of at least 0.02 mm3 in the absence of GA or nGA as diagnosed with OCT en face imaging OR Clinical diagnosis of early or early/intermediate stage AMD in one eye in the absence of nGA or GA and exudative AMD in the other eye OR clinical diagnosis of GA or nGA secondary to AMD that is at least the size of a large druse (125 microns in diameter; 0.05 mm2) and no greater than 7 disc areas (17 mm2) in at least one eye which has never been treated with anti-VEGF agents
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

* Subjects with exudative AMD in both eyes
* Eyes with evidence of non-proliferative and proliferative diabetic retinopathy.
* Presence of confounding ocular diagnosis such as myopia >6D, or other ocular conditions that may cause retinal pigment epithelium atrophy or exudative MNV
* Subjects currently or previously enrolled in other interventional clinical trials in which treatment was administered to the study eye.
* Previous vitrectomy or intravitreal injections in the study eye.
* Axial length measurement ≥ 26 mm.
* Subjects unable to give informed consent.
* Subjects who are unable to comply with imaging guidelines

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with intermediate AMD, Geographic Atrophy and nascent Geographic Atrophy and who have completed the BIRC-01 study
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-01-18 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in the Percentage of Choroidal Perfusion Deficits at 1 year compared to Baseline | 1-year and 2-year time points
  Compare the percentage of choroidal perfusion deficits as measured using automated algorithms

SECONDARY OUTCOMES:
Pre-existing and new sub-clinical Macular Neovascularization (MNV) | 1-year and 2-year time points
  Identify the number of abnormal new vessels arising from the Choroid at Baseline, 1-year and 2-year time points
Automated Drusen Volume measurements | 1-year and 2-year time points
  Compare the automated measurements of drusen volume using the Zeiss algorithm with manual measurements by trained readers
Automated Geography Atrophy measurements | 1-year and 2-year time points
  Compare the automated measurements of Geography Atrophy area using the Zeiss algorithm with manual measurements by trained readers
Choroidal Thickness (millimeters) | 1-year and 2-year time points
  Correlate Choroidal Thickness measurements (millimeters) with Age related Macular Degeneration (AMD) progression/Geographic Atrophy growth rates
Choroidal Vascularity Index (percentage) | 1-year and 2-year time points
  Correlate Choroidal Vascularity Index (percentage) with Age related Macular Degeneration (AMD) progression/Geographic Atrophy growth rates

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Waheed, MD, Principal Investigator — Boston Image Reading Center/Tufts Medical Center; Philip Rosenfield, MD, PhD, Principal Investigator — Bascom Palmer Eye Institute
Locations (5):
- United States (4):
  - University of California Los Angeles Doheny Eye Institute, Los Angeles, California
  - Bascom Palmer Eye Institue, Miami, Florida
  - New England Eye Center/Tufts Medical Center, Boston, Massachusetts
  - Vitreous Retina Macular Consultants of NY, New York, New York
- Melbourne University CERA, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided